CLINICAL TRIAL: NCT05869292
Title: Immediate Vs. Early Loading of Immediately Placed Bone Level Tapered Dental Implants
Brief Title: Immediate Vs. Early Loading of Immediately Placed Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Aleksa Markovic, Professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36/16
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Implant Complication; Implant
Keywords: immediate loading; Early loading; Marginal Bone Loss; Implant stability; Immediate implant placement
MeSH Terms: interventions — Immediate Dental Implant Loading; Control Groups

STUDY DESIGN:
Intervention Model Description: The study is design as a prospective, randomised, controlled clinical trial. Depending on number of extracted teeth patients will be randomly allocated into Test group in which immediate loading following surgical procedure will be conducted Control group in which early loading (six weeks postoperatively) will be performed.
Who Masked: Outcomes Assessor
Masking Description: Only investigators who will assess outcome including radiographic assessment, clinical outcomes and patients clinicians' satisfaction will be blinded all time. These investigators would not be familiar with group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test: Immediate implant loading (Experimental): Implants will be immediately following surgical procedure loaded with temporary restorations.
  Interventions: Device: Immediate implant loading
- Control: Early implant loading (Experimental): Implants will not be received prosthetic restoration, and will left with healing abutments (HA) for 6 weeks.
  Interventions: Device: Early implant loading

INTERVENTIONS:
Device: Immediate implant loading — Implants will be received immediately prosthetic restoration following surgical procedure.
  For the provisional restoration, an open tray impression technique will be used. Plaster models with scan bodies will be digitized by the laboratory scanner (3Shape E1, 3Shape, Kopenhagen, Denmark), and the virtual design of provisional restoration will be performed with 3D designing software (Exocad-Matera 2.3, Exocad, Darmstadt, Germany). Provisional restorations will be then created using polymethyl methacrylate (PMMA) (Telio®CAD, Ivoclar Vivadent, Schaan, Lichtenstein) and were drilled from PMMA blocks using the 5-axis milling machine (Zenotec Select, Wieland, Pforzheim, Germany). Screw-retained abutments for the prosthetic bridge will be chosen according to implant angulation and surrounding soft tissue height.
  At the end of the six-week healing period, definitive prosthetic restorations will be manufactured and delivered to the patients.
  Other Names: test group
  Arms: Test: Immediate implant loading
Device: Early implant loading — Implants won't receive immediately prosthetic restoration following surgical procedure and will be left only healing caps.
  At the end of the six-week healing period, definitive prosthetic restorations will be manufactured and delivered to the patients.
  Other Names: control group
  Arms: Control: Early implant loading

SUMMARY:
The study aims to compare implant stabilities between immediate and early loaded, immediately placed bone-level tapered dental implants in the upper jaw in the partial and total edentulous patients assessing marginal bone loss, oral health-related quality of life, and patient satisfaction within one, two and five years of follow-ups.

DETAILED DESCRIPTION:
The objectives of the study

The primary objective of this study will be to compare primary and secondary stability between immediate and early loaded, immediately placed bone-level tapered dental implants in the upper jaw in partial and total edentulous patients. The second objective will be marginal bone level changes and soft tissue changes such as keratinised tissue width and gingival thickness which will be assessed at one, two and five years postoperatively. The gained results will assess and compared within partial and total edentulous patients.

Additionally, the study also will be analyse functional and aesthetic outcomes as well as the possibility of the complication and its prevalences including (biological, mechanical, and procedure-related complications) comparing the their incidence between partial and total edentulous patients.

Materials and methods

The study is design as a prospective, randomised, controlled clinical trial which will be conducted at School of Dental Medicine in accordance with the Declaration of Helsinki (World Medical Association, 2013) and the CONSORT Statement.

Before the treatment procedure, after clinical examination patients will be divided into two groups:

1. Group A- patient requires on both sides one implant to be placed
2. Group B- patient requires full-arch reconstruction

Thereafter, in the both groups, patients will be randomly divided into two subgroups in which immediate loading (test group) or early loading (six week postoperatively) will be performed.

Surgical procedure

One hour before the surgery, antibiotic prophylaxis will be administered, and the patients should rins their mouths with 0.12% chlorhexidine solution for 1 minute preoperatively. The procedures will be performed under local anesthesia using 4% articaine, 1:100.000 epinephrine. A midcrestal incision will be made, and full-thickness will be elevated. Failing tooth or teeth will be extracted using periotomes, elevators, and forceps to preserve socket walls integrity. Extracted alveolus will be immediately prepared following by the epicrestal or subcrestal implant placement. If the gap between the implant surfaces and socket walls is wider than 2 mm, bovine-derived xenograft (Geistlich Bio-Oss®, Wolhusen, Switzerland) and collagen membrane (Geistlich Bio-Gide®, Wolhusen, Switzerland) will be placed. Healing screws (Institute Straumann AG, Basel, Switzerland; NC healing abutment ∅4.8 mm conical 5 mm and RC healing abutment ∅5 mm conical 6 mm) will be placed, and primary wound closure was achieved with 5-0 single resorbable sutures (AssuCryl Lactin, Pully-Lausanne, Switzerland). The presence of apical fenestration, cortical dehiscence, an apico-marginal defect, or the need for contour augmentation will also recorded in the patient study charts. Patients will be prescribed antibiotic therapy for the next five days (Amoxicillin with clavulonic acid, 1 g, twice a day, or, in case of allergy, Clindamycin, 0.6 g, three times a day).

2.3 Prosthetic protocol

Implants in subgroup marked as the test group will be immediately loaded with temporary restorations using S-R abutments (Institute Straumann AG, Basel, Switzerland) whereas the patients from the subgroup marked as control group wouldn't receive any kind of prosthetic restauration, and will left with healing abutments (HA).

For the provisional restoration, an open tray impression technique will be used. Plaster models with scan bodies will be digitized by the laboratory scanner (3Shape E1, 3Shape, Kopenhagen, Denmark), and the virtual design of provisional restoration will be performed with 3D designing software (Exocad-Matera 2.3, Exocad, Darmstadt, Germany). Provisional restorations will be then created using polymethyl methacrylate (PMMA) (Telio®CAD, Ivoclar Vivadent, Schaan, Lichtenstein) and were drilled from PMMA blocks using the 5-axis milling machine (Zenotec Select, Wieland, Pforzheim, Germany). Screw-retained abutments for the prosthetic bridge will be chosen according to implant angulation and surrounding soft tissue height.

At the end of the six-week healing period, definitive prosthetic restorations will be manufactured and delivered to the patients in both groups.

Data Collection and measurements

Implant stability, assessed as the primary study outcome, was measured using the Resonance Frequency Analysis (RFA) method with Osstell Mentor® (Osstell, Gothenburg, Sweden) (Fig. 7b) and Penguin® (PenguinRFA, Gothenburg, Sweden).

Marginal bone loss will be assessed as the difference between the postoperative and followed up years by means of CBCT measurements.

The distance between the implant shoulder and the crestal bone will be estimated as the shortest distance, using the same HA for each patient.

The results will be statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age;
2. systemically healthy;
3. periodontally healthy or with stable treated periodontitis and good oral hygiene (FMPS and FMBS ≤ 15%, measured at six sites per tooth)
4. Have maxillary dentition with one or multiple failing teeth
5. Have sufficient bone volume to immediately place implants
6. Non-smoker or light smoker

Exclusion Criteria:

1. An active or chronic disease that affects bone metabolism or wound healing (ASA III type);
2. Diminished mental capacities that could mitigate the ability to comply with the protocol;
3. History of maxillary augmentation; oral carcinoma or inflammatory changes;
4. History of head and neck radiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Implant stability | Change implant stability at 12 months
  Implant stability is measured using the Resonance Frequency Analysis (RFA) method with Osstell Mentor® (Osstell, Gothenburg, Sweden) and Penguin® (PenguinRFA, Gothenburg, Sweden). The result is expressed as ISQ values.
Implant stability | Change implant stability at 2 years
  Implant stability is measured using the Resonance Frequency Analysis (RFA) method with Osstell Mentor® (Osstell, Gothenburg, Sweden) and Penguin® (PenguinRFA, Gothenburg, Sweden). The result is expressed as ISQ values.
Implant stability | Change implant stability at 5 years
  Implant stability is measured using the Resonance Frequency Analysis (RFA) method with Osstell Mentor® (Osstell, Gothenburg, Sweden) and Penguin® (PenguinRFA, Gothenburg, Sweden). The result is expressed as ISQ values.

SECONDARY OUTCOMES:
Change of Marginal bone loss (MBL) | Change baseline marginal bone at 12 months
  MBL will be measured in millimetres as distance between the implant shoulder and the crestal bone postoperative and one, second, and five year postoperatively by using CBCT.
Change of Marginal bone loss (MBL) | Change baseline marginal bone at 2 years
  MBL will be measured in millimetres as distance between the implant shoulder and the crestal bone postoperative and one, second, and five year postoperatively by using CBCT.
Change of Marginal bone loss (MBL) | Change baseline marginal bone at 5 years
  MBL will be measured in millimetres as distance between the implant shoulder and the crestal bone postoperative and one, second, and five year postoperatively by using CBCT.
Change of keratinised tissue width (KTW) | Change baseline marginal bone at 12 months
  KTW will be measured in millimetres at the middle of the inserted implant as the distance between the free MM to a mucogingival junction (MGJ)
Change of keratinised tissue width (KTW) | Change baseline marginal bone at 2 years
  KTW will be measured in millimetres at the middle of the inserted implant as the distance between the free MM to a mucogingival junction (MGJ)
Change of keratinised tissue width (KTW) | Change baseline marginal bone at 5 years
  KTW will be measured in millimetres at the middle of the inserted implant as the distance between the free MM to a mucogingival junction (MGJ)

OTHER OUTCOMES:
Patient satisfaction | 12 moths postoperatively
  Patient will be recorded by using visual analog score (VAS). Patients will indicate their satisfaction relating to function, aesthetics, and discomfort/pain.
Patient satisfaction | 2 years postoperatively
  Patient will be recorded by using visual analog score (VAS). Patients will indicate their satisfaction relating to function, aesthetics, and discomfort/pain.
Patient satisfaction | 5 years postoperatively
  Patient will be recorded by using visual analog score (VAS). Patients will indicate their satisfaction relating to function, aesthetics, and discomfort/pain.
Pink aesthetic score (PES) | 12 months after implant loading
  A clinical photograph performed at 12 months examination, will be used for assessment.
  Seven variables of the implant supported crown will be evaluated vs. a contralateral natural tooth: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue color and texture. A 0-1-2 scoring system will be used, 0 being the lowest and 2 being the highest value.
Pink aesthetic score (PES) | 2 years after implant loading
  A clinical photograph performed at 2 years examination, will be used for assessment.
  Seven variables of the implant supported crown will be evaluated vs. a contralateral natural tooth: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue color and texture. A 0-1-2 scoring system will be used, 0 being the lowest and 2 being the highest value.
Pink aesthetic score (PES) | 5 years after implant loading
  A clinical photograph performed at 5 years examination, will be used for assessment.
  Seven variables of the implant supported crown will be evaluated vs. a contralateral natural tooth: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue color and texture. A 0-1-2 scoring system will be used, 0 being the lowest and 2 being the highest value.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksa Markovic, Professor, Study Director — School of Dental Medicine, University of Belgrade
Locations (1):
- School of Dental Medicine, Univeristy of Blegrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
The one and two years outcome will be statistically analysed and published in the journal which will be shared and available to public.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2022-2035
Access Criteria: The investigators will be shared analyzed outcomes and surgical procedure protocols

REFERENCES:
- [Background] Chambrone L, Shibli JA, Mercurio CE, Cardoso B, Preshaw PM. Efficacy of standard (SLA) and modified sandblasted and acid-etched (SLActive) dental implants in promoting immediate and/or early occlusal loading protocols: a systematic review of prospective studies. Clin Oral Implants Res. 2015 Apr;26(4):359-370. doi: 10.1111/clr.12347. Epub 2014 Feb 21. PMID 24814519
- [Background] Chung S, McCullagh A, Irinakis T. Immediate loading in the maxillary arch: evidence-based guidelines to improve success rates: a review. J Oral Implantol. 2011 Oct;37(5):610-21. doi: 10.1563/AAID-D-JOI-10-00058.1. PMID 22004059
- [Background] Del Fabbro M, Testori T, Kekovic V, Goker F, Tumedei M, Wang HL. A Systematic Review of Survival Rates of Osseointegrated Implants in Fully and Partially Edentulous Patients Following Immediate Loading. J Clin Med. 2019 Dec 4;8(12):2142. doi: 10.3390/jcm8122142. PMID 31817177
- [Background] Garcia-Sanchez R, Dopico J, Kalemaj Z, Buti J, Pardo Zamora G, Mardas N. Comparison of clinical outcomes of immediate versus delayed placement of dental implants: A systematic review and meta-analysis. Clin Oral Implants Res. 2022 Mar;33(3):231-277. doi: 10.1111/clr.13892. Epub 2022 Jan 28. PMID 35044012
- [Background] Ibrahim A, Chrcanovic BR. Dental Implants Inserted in Fresh Extraction Sockets versus Healed Sites: A Systematic Review and Meta-Analysis. Materials (Basel). 2021 Dec 20;14(24):7903. doi: 10.3390/ma14247903. PMID 34947493
- [Background] Markovic A, Misic T, Janjic B, Scepanovic M, Trifkovic B, Ilic B, Todorovic AM, Markovic J, Dard MM. Immediate Vs Early Loading of Bone Level Tapered Dental Implants With Hydrophilic Surface in Rehabilitation of Fully Edentulous Maxilla: Clinical and Patient Centered Outcomes. J Oral Implantol. 2022 Oct 1;48(5):358-369. doi: 10.1563/aaid-joi-D-21-00045. PMID 34937085